CLINICAL TRIAL: NCT07321301
Title: An Exploratory Clinical Study of CAR-T Cell Immunotherapy Using Polymer-lipid Particles to Deliver CAR1920 mRNA Targeting CD19/CD20 for Thetreatment of Relapsed/Refractory B-cell Lymphoma/Leukemia
Brief Title: Polymer-lipid Particle-delivered CAR1920 mRNA CAR-T Therapy for Relapsed/Refractory B-cell Lymphoma/Leukemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Daihong Liu (Other)
Responsible Party: Sponsor-Investigator, Daihong Liu, Dr., Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2025-727
Record Dates: First submitted 2025-12-22; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-10

CONDITIONS: B-cell Lymphoma Refractory
Keywords: consolidation therapy; B-cell Lymphoma Refractory; CAR-T; Lipid Nanoparticles; RNA Transport; Patient Safety

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with R/R B-Cell Lymphoma/Leukemia who accepted CD19/CD20 Dual-Targeting InViVoCAR-T (Experimental)
  Interventions: Drug: Polymer-Lipid Nanoparticle-Mediated Delivery of CD19/CD20 Dual-Targeting InViVoCAR1920 mRNA for CAR-T Cell Immunotherapy

INTERVENTIONS:
Drug: Polymer-Lipid Nanoparticle-Mediated Delivery of CD19/CD20 Dual-Targeting InViVoCAR1920 mRNA for CAR-T Cell Immunotherapy — Polymer-Lipid Nanoparticle-Mediated Delivery of CD19/CD20 Dual-Targeting InViVoCAR1920 mRNA for CAR-T Cell Immunotherapy in the Treatment of Patients with Relapsed/Refractory (R/R) B-Cell Lymphoma/Leukemia

SUMMARY:
The purpose of this study is to determine the efficacy and safety of the CAR-T cell immunotherapy utilizing polymer-lipid nanoparticles for delivering CD19/CD20 dual-targeting InViVoCAR1920 mRNA, for the first-line consolidation therapy of relapsed/refractory B-cell lymphoma/leukemia.

DETAILED DESCRIPTION:
Since 2010, Chimeric Antigen Receptor T-Cell Immunotherapy (CAR-T Cell Immunotherapy) has demonstrated excellent targeting, cytotoxicity, and durability in tumor treatment, achieving well-recognized clinical efficacy in hematological malignancies. CAR-T Cell Immunotherapy refers to a technique that uses genetic modification to introduce genetic material encoding a specific antigen-recognition domain and T-cell activation signals into T cells. These engineered T cells are activated by direct binding to specific antigens on the surface of tumor cells, directly killing tumor cells through the release of perforin, granzyme B, etc. Simultaneously, they recruit endogenous immune cells in the human body to eliminate tumor cells by secreting cytokines, thereby achieving tumor treatment. Furthermore, they can form memory T cells to establish a specific and long-term anti-tumor mechanism.CD19 and CD20 are specific markers of B-cell malignancies, widely expressed in various B-cell malignant tumors. However, single-antigen targeting is prone to inducing antigen escape, as tumor cells often evade recognition and attack by CAR-T cells by losing or downregulating the expression of a single target antigen. Nevertheless, it is relatively difficult for tumor cells to alter the expression of two antigens simultaneously. For example, 70% of patients who relapse after CD19 CAR-T therapy exhibit loss of CD19 expression, a population that can be covered by CD20 CAR-T therapy. However, the efficacy of single-agent therapy is still limited by antigen heterogeneity. Dual-target CAR-T cells simultaneously target CD19 and CD20 antigens. Even if tumor cells escape via one antigen, they can still exert cytotoxic effects through recognition of the other antigen, thereby significantly reducing the risk of antigen escape, improving tumor clearance efficiency, and lowering the recurrence rate.Lipid Nanoparticles (LNPs) are composed of cationic lipids, helper lipids, cholesterol, and polyethylene glycol (PEG)-modified lipids. They can efficiently encapsulate mRNA to form stable nanoscale particle structures, effectively protecting mRNA from degradation by nucleases in the body. Through interaction with the cell surface, LNPs can precisely deliver mRNA into T cells, enabling transient expression of CAR proteins and in situ generation of CAR-T cells. This technology eliminates the need for ex vivo cell manipulation, significantly shortening the treatment cycle and allowing patients to receive therapy more quickly. Meanwhile, it avoids the potential T-cell exhaustion that may occur during ex vivo T-cell expansion, improving the yield of effective therapeutic products.

ELIGIBILITY:
Inclusion Criteria:

1. Has voluntarily given informed consent, signed the informed consent form, and is willing and able to comply with the scheduled visits, study treatment, laboratory tests, imaging examinations, and other necessary trial procedures as required in the protocol;
2. Patients with relapsed/refractory (R/R) B-cell lymphoma/leukemia confirmed by histopathology, cytogenetics, molecular biology, clinical judgment, medical history, and other assessment methods in accordance with the WHO 2016 classification criteria, who have experienced disease progression under standard treatment regimens, are intolerant to standard treatment regimens, or lack effective standard treatment options;
3. Must meet the following criteria for R/R B-cell malignant tumors:

(1) B-cell tumors include 3 categories:

* B-cell acute lymphoblastic leukemia (B-ALL);

  ② Indolent B-cell lymphomas, including chronic lymphocytic leukemia (CLL), follicular lymphoma (FL), marginal zone lymphoma (MZL), lymphoplasmacytic lymphoma (LPL), hairy cell leukemia (HCL), etc.;

  ③ Aggressive B-cell lymphomas, including diffuse large B-cell lymphoma (DLBCL), Burkitt lymphoma (BL), mantle cell lymphoma (MCL); (2) R/R B-ALL (meeting any 1 of the 4 criteria below):
* Relapse within 6 months after the first complete response (CR);

  * Primary refractory patients who failed to achieve CR after 2 cycles of standard chemotherapy;

    * Failure to achieve CR or relapse after first-line or multi-line salvage chemotherapy; ④ Relapse after hematopoietic stem cell transplantation (HSCT); (3) R/R B-cell lymphoma (meeting any 1 of the first 4 criteria below plus criterion 5):
* Tumor reduction < 50% or disease progression after 4 courses of standardized chemotherapy per standard regimens;

  * Relapse within 6 months after achieving CR with standard chemotherapy;

    * ≥ 2 relapses after CR;

      * Relapse after HSCT; ⑤ Adequate prior treatment received, including at least anti-CD20 monoclonal antibody and anthracycline-containing combination chemotherapy regimens; 4. Aged 18-85 years (inclusive), male or female; 5. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2; 6. Expected survival > 14 days from the date of signing the informed consent form; 7. Hemoglobin (HGB) ≥ 60 g/L (transfusion allowed); 8. Absolute neutrophil count (ANC) ≥ 1,000/μl and platelet count ≥ 45,000/μl in peripheral blood (transfusion allowed); 9. Hepatic, renal, cardiac, and pulmonary functions meeting the following requirements:

        1. Total Bilirubin (TBIL) ≤ 1.5 × Upper Limits of Normal (ULN), excluding subjects with Gilbert's syndrome;
        2. Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST) ≤ 2.5 × ULN;
        3. Serum Creatinine (Cr) ≤ 1.5 × ULN or Creatinine Clearance Rate (CCr) ≥ 60 mL/min (CCr estimated by the Cockcroft-Gault formula);
        4. Left Ventricular Ejection Fraction (LVEF) ≥ 50%; echocardiogram (ECHO) confirms no clinically significant severe pericardial effusion or severe arrhythmia;
        5. Baseline transcutaneous oxygen saturation > 90% under room air;
        6. No clinically significant severe pleural effusion; 10. Subjects with pregnancy plans must agree to use contraceptive measures from before study enrollment until 6 months after the end of the study;

Exclusion Criteria:

1. Previous receipt of any form of chimeric antigen receptor (CAR) cell therapy or other genetically modified T-cell therapies;
2. History of severe immediate-type hypersensitivity reactions to commonly used drugs such as aminoglycoside antibiotics;
3. Known history of Human Immunodeficiency Virus (HIV) infection, active Hepatitis B Virus (HBV) infection, or any uncontrolled active systemic infection requiring intravenous antibiotics (active HBV infection is defined as meeting all three of the following criteria: a. HBV DNA quantitation ≥ 2000 IU/ml; b. ALT ≥ 2 × Upper Limits of Normal (ULN); c. Exclusion of hepatitis caused by other factors such as the disease itself or medications. If a patient was diagnosed with active HBV infection initially and converted to inactive HBV infection after anti-HBV treatment, they may be included in this study with adequate ongoing anti-HBV treatment);
4. Hepatic or renal impairment unrelated to hematologic malignancies (e.g., lymphoma): ALT > 3 × ULN, AST > 3 × ULN, TBIL > 2 × ULN, or serum creatinine clearance < 30 mL/min;
5. History of myocardial infarction, cardiac angioplasty, coronary artery stenting, unstable angina pectoris, active arrhythmia, or other clinically significant cardiovascular diseases within 12 months prior to enrollment;
6. Other severe medical conditions that may affect the study (e.g., poorly controlled diabetes mellitus, gastric ulcer, other severe cardiorespiratory diseases, concurrent severe autoimmune diseases or congenital immunodeficiencies, uncontrolled severe infections, etc.), as well as other diseases with a high risk of condition deterioration; patients who received allogeneic hematopoietic stem cell transplantation (allo-HSCT) and still have acute graft-versus-host disease (GVHD) 1 month after discontinuing immunosuppressants. The decision is at the investigator's discretion;
7. History of severe immediate-type hypersensitivity reactions to any specific drugs required in this study; or history of severe hypersensitivity to biological products (including antibiotics);
8. Female subjects who are pregnant or lactating (due to potential risks of treatment to the fetus or infant);
9. Subjects judged by the investigator to be unable to complete all scheduled visits, investigations, or diagnostic and therapeutic procedures required by the study protocol (including medium- and long-term follow-up visits), those with poor willingness to participate, those who are unwilling to join or fully cooperate with the study arrangements, or those with insufficient compliance of the subject and their family members. The decision is at the investigator's discretion;
10. Concurrent progressive malignant tumors of other types; or a history of other malignant tumors, except for non-melanoma skin cancers and carcinoma in situ (e.g., of the cervix, bladder, or breast). Subjects with a history of other malignant tumors are ineligible unless they have been disease-free and not received any form of anti-tumor treatment for at least 3 consecutive years;
11. History of live vaccine vaccination within 6 weeks prior to the start of the conditioning regimen;
12. Receipt of major surgical procedures (excluding lymph node biopsy) within the past 14 days, or anticipated need for major surgery during the treatment period;
13. Other severe physical or mental illnesses or laboratory abnormalities that may increase the risk of study participation or interfere with study results, as well as patients deemed unsuitable for participation by the investigator.

Ages: 14 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
the safety and maximum tolerated dose of CAR-T cell immunotherapy mediated by polymer-lipid nanoparticles delivering CD19/CD20 dual-targeting InViVoCAR1920 mRNA in patients with relapsed/refractory B-cell lymphoma/leukemia | 3 months after treatment

SECONDARY OUTCOMES:
30-day response rate | 30 days
  30-day response rate refers to the proportion of patients who achieve complete or partial response from the start of treatment.
90-day response rate | 90 days
  90-day response rate refers to the proportion of patients who achieve complete or partial response 90 days after the start of treatment.
overall survival (OS) | 6 months after treatment
  Overall survival (OS) refers to the time from the start of treatment to the death of the patient for any reason
progression free survival (PFS) | 6 months after treatment
  Progression free survival (PFS) refers to the time from treatment to the first myeloma progression or death of the patient for any reason.
time to progression (TTP) | 6 months after treatment
  Time to progression (TTP) refers to the time from treatment to the first myeloma progression.
disease free survival (DFS) | 3 months after treatment
  Disease free survival (DFS) refers to the time from treatment to the first myeloma recurrence.
duration of response (DOR) | 6 months after treatment
  Duration of Response (DOR) refers to the time from the first assessment of a myeloma as a complete or partial response to the first assessment of PD (Progressive Disease) or death from any cause.
event free survival (EFS) | 6 months after treatment
  Event Free Survival (EFS) is a commonly used endpoint indicator in clinical trials to evaluate the survival time of patients without any adverse events during a specific time period. These adverse events include but are not limited to disease progression, death, treatment plan changes, and the occurrence of serious side effects.
recurrence rate | 3 months after treatment
  The recurrence rate refers to the proportion of patients with lymphoma recurrence after treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No